CLINICAL TRIAL: NCT04044508
Title: Odified Ketogenic Diet in Patients With McArdle Disease Part B - a Placebo-controlled, Cross-over Study
Brief Title: Modified Ketogenic Diet in Patients With McArdle Disease Part B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Nicoline Løkken, MD, Research fellow, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-18013022-B
Record Dates: First submitted 2018-12-12; First posted 2019-08-05 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: McArdle Disease
MeSH Terms: conditions — Glycogen Storage Disease Type V | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized, blind, placebo-controlled, cross over study
Who Masked: Participant, Investigator
Masking Description: Disguise products (Oral supplements: Nutricia 'ketocal' (intervention) or Nutricia 'fortini' (placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional diet (Active Comparator): A modified ketogenic diet (with the composition found in the pilot study, 75%fat, 15% protein, 10% carbohydrates)
  Interventions: Dietary Supplement: Ketocal 4:1 liquid Nutricia (intervention)
- Placebo diet (Placebo Comparator): A placebo diet (over 100 g of carbohydrates per day)
  Interventions: Dietary Supplement: Fortini multifibre Nutrica (placebo)

INTERVENTIONS:
Dietary Supplement: Ketocal 4:1 liquid Nutricia (intervention) — Modified ketogenic diet
  Arms: Interventional diet
Dietary Supplement: Fortini multifibre Nutrica (placebo) — Placebo diet
  Arms: Placebo diet

SUMMARY:
McArdle disease, glycogen storage disease type V, is a rare metabolic disease. Affected individuals are unable to utilize sugar stored as glycogen in muscle. Investigators hypothesize that a modified ketogenic diet could be a potential treatment option, by providing ketones as alternative fuel substrates for working muscle.

This blinded, placebo-controlled, cross-over study will investigate the potential effects of an optimal modified ketogenic diet found in part A (75% fat, 15%protein, 10%carbohydrates) in patients with McArdle disease compared with a healthy balanced placebo diet (>100grams of carbohydrates per day).

DETAILED DESCRIPTION:
A blinded randomized, placebo-controlled, cross-over study to investigate the effects of a modified ketogenic diet in patients with McArdle disease.

McArdle disease, glycogen storage disease type V, is a rare metabolic disease caused by mutations in the PYGM gene resulting in absence of the enzyme muscle phosphorylase. Affected individuals are unable to utilize sugar stored as glycogen in muscle, leading to exercise intolerance, exercise-induced muscle pain, contractures and rhabdomyolysis. Currently, there are no satisfactory treatment options for McArdle disease. Ketones are feasible fuel alternatives to muscle glycogen when muscle glycogenolysis is blocked as in McArdle disease. A key element of alleviating symptoms in McArdle disease is to provide alternative fuels for energy metabolism. Ketosis can potentially provide alternative fuel substrates by provision of endogenous ketone bodies (KBs) which are desirable fuels for skeletal muscle and brain. Ketosis can be reached by fasting and can be induced by adhering to a modified ketogenic diet, which entails a high-fat, low-carbohydrate diet, which simulates the metabolic effects of fasting.

The study design is a placebo-controlled, blind, cross over design. The study will be carried out at two sites: CNMC (Copenhagen), NHNN (London). Subjects will be randomized 1:1 to receive either a modified ketogenic diet (75% fat, 15%protein, 10% carbohydrates) or a placebo diet (>100grams of carbohydrates per day) first. Subjects will follow the diet for 4 weeks, followed by 2-4 weeks wash-out, followed by 4 weeks on the opposite diet. During the 10-12 weeks trial period, subjects will visit the trial site in London on five occasions. Effects of the diet will be evaluated by improvement in exercise capacity during submaximal exercise test on a cycle ergometer. Subjective improvements will be evaluated by questionnaires and a dietary diary.

If the diet improves exercise capacity, it will provide a safe and cheap treatment option that may lead to reduced risk of muscle injury and enhance quality of life in patients with McArdle disease.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed GSDV
* Patient is willing and able to provide written informed consent prior to participation.
* Patient is ambulatory.
* Women in fertile age must be willing to practice the following medically acceptable methods of birth control

Exclusion Criteria:

* Patient has any prior or current medical conditions that, in the judgment of the Investigator, would prevent the patient from safely participating in and/or completing all study requirements.
* Pregnancy or breastfeeding
* Patient does not have the cognitive capacity to understand/comprehend and complete all study assessments
* Patients with porphyria or disorders of fat metabolism (primary carnitine deficiency, carnitine palmitoyltransferase I or II, β-oxidation defects etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-03 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in mean heart rate | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Change in mean heart rate (bpm) during constant load cycling exercise (30 minute submaximal cycle test). Heart rate will be measured every minute during the cycle test at all visits.

SECONDARY OUTCOMES:
Compliance | up 12 weeks
  Daily dietary diary
Change in Indirect calorimetry | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Oxidation rates measured via indirect calorimetry during constant load cycling Measured at visit 1-4.
Change in self-rated daily function scores | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Modified SF-36 questionnaire
Change in self-rated fatigue | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Fatigue Severity Scale score
Change in blood ketones | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Ketone bodies in the blood (hydroxybutyrate+acetoacetate umol/L).
Change in perceived exertion | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Borg scale (scale from 6-20). During the constant load cyclinging test, subjects will be asked every minute during.
Change in ammonia | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Blood Ammonia (umol/L). Will be measured 5 times during the cycle test at visit 1-4.
Change in insulin | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Blood Insulin (pmol/l). Will be measured 6 times during the cycle test at visit 1-4.
Change in Adrenalin | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Blood Adrenalin (pg/mL) Will be measured 6 times during the cycle test at visit 1-4.
Change in glucagon | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Blood Glucagon (pmol/L). Will be measured 4 times during the cycle test at visit 1-4.
Change in maximal oxygen capacity | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  (VO2max, mL oxgen per minute) after the 30 minutes submaximal exercise test, the workload will be increased in a step vise manner to maximum.
Change in maximal work load | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Work load (watts) after the 30 minutes submaximal exercise test, the workload will be increased in a step vise manner to maximum.
Change in free fatty acids | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Blood Free fatty acids (umol/L). Will be measured 6 times during the cycle test at visit 1-4.
Change in lactate | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Blood Lactate (mM). Will be measured 6 times during the cycle test at visit 1-4.
Change in glucose | At Visit 1 (baseline), Visit 2 (4 weeks), Visit 3 (8 weeks), and Visit 4 (12 weeks)
  Blood glucose (mM). Will be measured 6 times during the cycle test at visit 1-4.

CONTACTS AND LOCATIONS:
Locations (2):
- Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Denmark
- National Hospital for Neurology and neurosurgery, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lokken N, Nielsen MR, Stemmerik MG, Ellerton C, Revsbech KL, Macrae M, Slipsager A, Krett B, Beha GH, Emanuelsson F, van Hall G, Quinlivan R, Vissing J. Can a modified ketogenic diet be a nutritional strategy for patients with McArdle disease? Results from a randomized, single-blind, placebo-controlled, cross-over study. Clin Nutr. 2023 Nov;42(11):2124-2137. doi: 10.1016/j.clnu.2023.09.006. Epub 2023 Sep 20. PMID 37769369